CLINICAL TRIAL: NCT03160469
Title: Prospective Study Of The Procedure-less Intra-gastric Elipse Balloon: Is It Effective & Safe?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amiri Hospital (Other Government)
Responsible Party: Principal Investigator, Saud AL-Subaie, MD , Specialist surgeon, Amiri Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AmiriH
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Obese
Keywords: obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This is a prospective pilot study of 48 patients underwent Elipse balloon insertion by the same surgeon at Faisal polyclinics in Kuwait city during six months period from July 2016 to January 2017. Ethical approval was obtained from the Ministry of Health in Kuwait & national ethics committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elipse capsule insertion group (Experimental): All patient who inserted elipse capsule in single clinic
  Interventions: Device: intragastric Elipse Device

INTERVENTIONS:
Device: intragastric Elipse Device — Obesity prevalence is increasing worldwide, and Kuwait is currently considered to be the country with the most obese population1. Accordingly, standardization of the weight loss procedures has been made according to the Body Mass Index (BMI), keeping the more advanced surgeries for class II obesity (BMI 35- 39.9) and above, with consideration of other factors like, for example, obesity-related comorbidities. For those patients whom considered in the category of overweight (BMI = 25- 29.9) & class I obesity (BMI 30- 34.9), after failure of diet attempts, the weight loss options are limited. Of the highly requested options are the various types of intra-gastric balloons. Conventional endoscopic gastric balloons have proven to be safe and effective, with Excess Weight Loss (%EWL) of 25-50%2. A new swallowable gastric balloon, named Elipse, has been launched recently in Kuwait and became highly popular due to its unique concept of being "procedure-less".

SUMMARY:
a prospective intragastric elipse balloon effect on weight loss for certain BMI. this study also proposed to assess the safety of the elipse balloon

DETAILED DESCRIPTION:
Obesity prevalence is increasing worldwide, and Kuwait is currently considered to be the country with the most obese population1. Accordingly, standardization of the weight loss procedures has been made according to the Body Mass Index (BMI), keeping the more advanced surgeries for class II obesity (BMI 35- 39.9) and above, with consideration of other factors like, for example, obesity-related comorbidities. For those patients whom considered in the category of overweight (BMI = 25- 29.9) & class I obesity (BMI 30- 34.9), after failure of diet attempts, the weight loss options are limited. Of the highly requested options are the various types of intra-gastric balloons. Conventional endoscopic gastric balloons have proven to be safe and effective, with Excess Weight Loss (%EWL) of 25-50%2. A new swallowable gastric balloon, named Elipse, has been launched recently in Kuwait and became highly popular due to its unique concept of being "procedure-less".

Elipse is a weight loss device that does not require anesthesia, endoscopy, or surgery in its "way in" or "way out". It's designed to be a swallowable capsule that is converted to a balloon in the stomach after filling it with a PH-titrated fluid through its connected catheter. It works by restricting the stomach and, as a result, weight loss is achieved by decreasing the overall food quantity intake. Four months later, part of the balloon patch side is shed-off and the fluid is expelled in the stomach in a gradual manner. Later, the fluid and the thin paper-like wall of the balloon pass through the gastrointestinal tract until excreted.

This prospective study aims to observe the efficacy & safety of the procedure-less intra-gastric Elipse balloon as a tool aiding in weight loss applied to all patients in our clinic who fulfill the criteria & underwent insertion procedure by one surgeon. In this paper we share our experience regarding this new type of balloon, since Kuwait is one of the first countries to start official practice with this new device and data in literature is still lacking.

This is a prospective pilot study of 48 patients underwent Elipse balloon insertion by the same surgeon at Faisal polyclinics in Kuwait city during six months period from July 2016 to January 2017. After insertion, the patients were followed for a period of four months until the expected day of excretion. Weight, BMI, & waist circumference were calculated once pre-insertion and at 1,2, and 4 months post-insertion in the clinic. Patients were also encouraged to send their body composition data through email using electronic scale at home in weekly basis. All the data regarding any difficulties or adverse events during the procedure were recorded. At the last visit, a simple questionnaire was handed to the patients to address the commitment to peri and post procedural instructions, symptoms & their severity encountered after insertion and excretion, overall costs spent, and patient satisfaction. Ethical approval was obtained from the Ministry of Health in Kuwait & national ethics committee.

ELIGIBILITY:
Inclusion Criteria:

all patients underwent elipse insertion from July 2016 to January 2017with:

* BMI 27-40
* Age 18-65
* Failed multiple diet attemps
* Motivated with realistic weight loss expectations, ready and committed to follow a physician-guided weight-loss program.

Exclusion Criteria:

* Patients with psychologically-driven eating disorders (e.g. binge eating, bulimia, etc.)
* Patients with a history of abdominal and/or pelvic surgery EXCLUDING only ONE of the following surgeries that was performed at least 12 months prior to the Elipse™ Treatment: cesarean section, diagnostic laparoscopy, laparoscopic appendectomy, laparoscopic cholecystectomy.
* Patient has had previous bariatric or gastric surgery.
* Patient has a history of acute pancreatitis.
* Patient has a history of small bowel obstructions.
* Patient has history of/or signs and/or symptoms of esophageal, gastric, or duodenal disease including but not limited to hiatal hernias >2 centimeter (cm), inflammatory diseases, cancer, and varices.
* Patients with an abnormal swallowing mechanism.
* Patients with a history of cancer, inflammatory disease, bleeding or other disorder of the gastrointestinal (GI) tract.
* Women who are pregnant or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
weight loss | 4 months
  weight loss

SECONDARY OUTCOMES:
symptoms & its severity | 4 months
  nausea , vomiting, abdominal pain
patient satisfaction | 4 months
  overall patient satisfaction:
  patients were given a short questionnaire with a scale from (0 - 10) for each: ease of the procedure, symptoms and severity, satisfaction with the results, & the overall costs.
overall cost | 4 months
  overall cost spent for this procedure

IPD SHARING:
Plan to Share IPD: Yes
This is a study for publication in International surgical journal to be shared by all clinicians using this device